CLINICAL TRIAL: NCT05516576
Title: Endoscopic Sutured Gastroplasty with Endomina® Device Versus Standard of Care in Patients with Type 2 Diabetes and Class I Obesity: a Multi-center, Randomized Controlled Trial
Acronym: ESTIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Endo Tools Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-2019-002
Record Dates: First submitted 2022-07-15; First posted 2022-08-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- endoscopic gastroplasty with endomina® (Experimental)
  Interventions: Device: endomina®
- control (No Intervention)

INTERVENTIONS:
Device: endomina® — Endoscopic gastroplasty
  Arms: endoscopic gastroplasty with endomina®

SUMMARY:
The primary objective of this study is to assess the efficacy of endoscopic gastric reduction with the endomina® device, in combination with standard of care, compared to standard of care alone, on the remission of diabetes 24 months after surgery, in patients with type-2 diabetes and class I obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years;
* Recently diagnosed Type 2 Diabetes (<= 10 years):
* HbA1c < 9%:
* Under non-insulin anti-diabetic treatment, i.e., metformin, sulfonylurea, glinide, DPP4i, GLP1-RA, SGLT2i, alone or in combination
* Anti-diabetic therapy stable during the last 3 months before inclusion
* BMI between 30-34.9 kg/m² with adaptation for Asian population 27.5-32.5kg/m²
* Must be able to comply with all study requirements for the duration of the study as outlined in the protocol (including compliance to randomization treatment, dietary follow up, visits schedule and all study specific procedures);
* Must be able to understand and be willing to provide written informed consent.

Exclusion Criteria:

* Contra-indication to the use of endomina® and TAPES according to their Instruction for Use (IFU).
* Type I diabetes characterized by C peptide <0.2 nmol/l or presence of anti-GAD, anti IA2, anti-ZNT8
* Unstable diabetic retinopathy
* Severe kidney (stage 4-5), hepatic (child B and C cirrhosis), pulmonary disease or cancer (cancer in the past 5 years);
* Short-term prognosis due to a proven serious comorbidity including severe macrovascular complications and / or a limited life expectancy (<5 years)
* Contra-indication to endoscopic gastroplasty (...)
* Impending gastric surgery 60 days post intervention;
* Participant involved in another interventional clinical study
* Patients having alcoholic or drug addiction;
* Patients having a severe mental illness such as psychosis, bipolar disorders, severe, current depression or eating disorder such as bulimia nervosa or binge eating disorder;
* Person deprived of liberty by judicial order
* Person under guardianship or curatorship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Remission of diabetes after endoscopic gastroplasty with endomina, in patients with type-2 diabetes and class I obesity | 24 months
  Remission is defined as HbA1c < 6.5% without antidiabetic drug for at least 3 months

CONTACTS AND LOCATIONS:
Overall Officials: A-L BOREL, MD PHD, Principal Investigator — University Grenoble Hospital
Locations (1):
- Chu Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided